CLINICAL TRIAL: NCT02810561
Title: Time Course and the Significance of Troponin Leaks in Emergency Department Patients Presenting With Supraventricular Tachycardia (SVT)
Brief Title: Troponin Leaks in Emergency Department Patients Presenting With Supraventricular Tachycardia (SVT)
Status: Completed | Type: Observational
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Other Study IDs: LH01
Record Dates: First submitted 2016-04-26; First posted 2016-06-23 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Supraventricular Tachycardia
Keywords: Troponin
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No intervention was completed with this study.

SUMMARY:
The goal of this study is twofold. First the investigators would like to determine the trajectory of troponin leaks; if it can be shown that the participants who have only minimal elevations of their repeat troponin universally decrease on the 3rd level then future patients may see significantly improved length of stay. Second, given conflicting results in the literature, the investigators would like to determine if elevated troponin levels correlate to later cardiovascular complications. These complications will be defined as Death, Myocardial Infarction, Cardiovascular intervention (such as coronary artery stenting or bypass). As the investigator is a single hospital system in this county it is uniquely positioned to be able to review this retrospectively.

DETAILED DESCRIPTION:
The investigators therefore propose retrospectively studying participants diagnosed with Supraventricular Tachycardia who had troponin(s) checked in the ED between January 1, 2012 and May 31, 2016 to allow a minimum of a year follow-up for our combined endpoint. The investigators will record the participants troponin value(s) in addition to the age, sex, race, heart rate, creatinine value. The investigators will compare the participants with positive troponins (and hopefully participants with strongly positive troponins) with those who are negative for troponin for presence of the combined end point via chart review.

ELIGIBILITY:
Inclusion Criteria:

* Supraventricular Tachycardia with troponin elevation

Exclusion Criteria:

* Other cardiac arrhythmias or conditions with increased troponin

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to the Emergency Department with Supraventricular Tachycardia and elevated troponin. All sexs, races and ages will be included.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Troponin-I Level | 6 hours after initial EKG
  Measured in ng/ml

SECONDARY OUTCOMES:
Death/ Need for Cardiac Stent Placement or Coronary Bypass Artery Graft | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hysell, MD, Principal Investigator — Lakeland Health Emergency Department

IPD SHARING:
Plan to Share IPD: Undecided